CLINICAL TRIAL: NCT04261777
Title: A Confirmatory, Prospective, Open-label, Single-arm, Reader-blinded Multi-centre Phase 3 Study to Assess the Diagnostic Accuracy of Ferumoxtran-10-enhanced Magnetic Resonance Imaging (MRI) and Unenhanced MRI in Reference to Histopathology in Newly-diagnosed Prostate Cancer (PCA) Patients, Scheduled for Radical Prostatectomy (RP) With Extended Pelvic Lymph Node Dissection (ePLND).
Brief Title: Ferumoxtran-10-enhanced MRI in Prostate Cancer Patients
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was closed prematurely in order to finalise it under EU directive 2001/20/EC, without transitioning to EU-CTR, and avoiding unnecessary delay of the marketing authorisation application.
Sponsor: Saving Patients' Lives Medical B.V. (Industry)
Collaborators: ABX-CRO advanced pharmaceutical services Forschungsgesellschaft m.b.H. (Unknown); b.e.imaging GmbH (Unknown); Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SPL-01-001
Record Dates: First submitted 2020-01-27; First posted 2020-02-10 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Prostate Cancer; Metastasis; Prostatectomy
Keywords: SPL-01-001; ePLND; MRI; USPIO; MR lymphography; Ferrotran; Ultra-small superparamagnetic iron oxide; Nanoparticles
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasm Metastasis | interventions — ferumoxtran-10

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- SPL-01-001 (Experimental)
  Interventions: Drug: Ferrotran® (Ferumoxtran-10)

INTERVENTIONS:
Drug: Ferrotran® (Ferumoxtran-10) — Ferrotran® in a dose of 0.13 mL/kg body weight of the reconstituted freeze-dried preparation (i.e. 2.6 mgFe/kg body weight). The recommended dose should be diluted in 100 mL of NaCl 9 mg/mL (0.9%) solution for injection/infusion prior to administration via the infusion filter as a slow intravenous infusion over 30 minutes (at a maximum rate of 4 mL/min).
  Ferrotran® will be administered once to each patient. Histologically confirmed diagnosis and pre-operative staging are performed prior to the study as part of standard care. Surgery (RP with ePLND) and sampling of tissue specimens is performed after the Ferrotran®-enhanced MRI as part of standard care.
  Other Names: Ferrotran Lyophilisate

SUMMARY:
This will be a confirmatory, prospective, open-label, single-arm, reader-blinded, multi-centre phase 3 study to assess the diagnostic accuracy and safety of Ferrotran®-enhanced MRI in comparison to unenhanced MRI in the detection of pelvic lymph node metastases in newly-diagnosed adult patients with prostate cancer and an intermediate to high risk for lymph node metastases, based on the D'Amico criteria.

DETAILED DESCRIPTION:
Potential patients for this study will be recruited by up to 15 centres specialised in prostate cancer. Study sites will be interdisciplinary, consisting of a uro-oncology sub-site, and a radiology sub-site with high-quality MRI, surgery and pathology. Study visits will be typically conducted at the recruiting sub-site, or as institutionally appropriate. Treatment visits for patients will be performed in the collaborating sub-site. Patients will be invited for study participation by the investigators in the context of specialised clinics. Interested patients will be provided with an information sheet and will undergo a detailed informed consent procedure prior to any study procedures. Recruitment will be continued until a sufficient number of patients have undergone Ferrotran® imaging and histopathological evaluation.

To compensate for an expected drop-out rate of 15% to 20%, recruitment will only be stopped as soon as at least 69 evaluable positive (patients positive) and at least 104 evaluable negative (patients negative) patients are available for analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily given and written informed consent.
2. Male ≥18 years of age.
3. Histologically newly-confirmed adenocarcinoma of the prostate.
4. Medium to high risk for lymph node metastasis, defined by either:

   1. PSA ≥10 ng/mL or
   2. Gleason-Score ≥7 or
   3. Stage cT2b or cT2c or T3 or T4
5. Patients scheduled for radical prostatectomy (RP) with extended lymph node dissection (ePLND) between Day 7 and Day 42 after Ferrotran®-enhanced MRI.
6. Consent to practice contraception until end of study, including female partners of childbearing potential. Effective contraceptive measures include hormonal oral, injected or implanted female contraceptives, male condom, vaginal diaphragm, cervical cap, intrauterine device.

Exclusion Criteria:

1. Any contraindication to MRI, as per standard criteria.
2. Any radiation therapy or systemic antiproliferative (chemo-, immuno, or hormonal) therapy for prostate cancer (Lupron, Taxotere, Casodex, Eulexin, Zoladex, etc.) prior to screening and until after post-surgery FUP MRI.
3. Known hypersensitivity to Ferrotran® or its components such as dextran.
4. Known hypersensitivity to other parenteral iron products.
5. Acute allergy, including drug allergies and allergic asthma.
6. Evidence of iron overload or disturbances in the utilisation of iron (e.g., haemochromatosis, haemosiderosis, chronic haemolytic anaemia with frequent blood transfusions).
7. Presence of liver dysfunction.
8. Any other investigational medicinal product within 30 days prior to receiving study medication until end of study visit.
9. Simultaneous participation in any other clinical trial.
10. Abnormal safety laboratory values at screening or baseline that are assessed by the principal investigator as clinically relevant.
11. Patients not able to declare meaningful informed consent on their own (e.g. with legal guardian for mental disorders), or other vulnerable patients (e.g. under arrest).
12. Patients with acute SARS-CoV-2 infection

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — male with prostate cancer
Enrollment: 172 (Actual)
Dates: Start 2020-05-27 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-01-15 (Actual)

PRIMARY OUTCOMES:
Lymph node metastases will be detected by MRI scan (Ferumoxtran-10-enhanced and unenhanced). | up to day 42
  True positive fraction and false positive fraction of identified tumour tissue in pelvic lymph nodes will be analysed by histopathology as established reference method.

SECONDARY OUTCOMES:
Number and regions of lymph node metastases present in the follow-up MRI in comparison to pre-surgery MRI (unenhanced and Ferrotran®-enhanced). | up to day 105
Frequency of occurrence and severity of abnormal findings in safety investigations (physical examination, vital signs, 12-lead ECG, clinical laboratory, concomitant medication, adverse events) | day 0 - day 105
Percentage of subjects for whom the patient management plan would be changed based on the Ferrotran®-enhanced MRI. | up to day 105

CONTACTS AND LOCATIONS:
Locations (15):
- Universitair Ziekenhuis Ghent, Ghent, Belgium
- Germany (10):
  - Charité - Universitätsklinikum Berlin, Berlin, State of Berlin
  - Vivantes Klinikum Am Urban, Berlin
  - Universitätsklinikum Bonn, Bonn
  - Universitätsklinikum Köln, Cologne
  - Universitätsklinikum Carl Gustav Carus, Dresden
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - Universitätsklinikum Essen, Essen
  - Universitätsklinikum Leipzig, Leipzig
  - Universitätsklinikum Schleswig-Holstein Lübeck, Lübeck
  - Universitätsmedizin Mannheim Medizinische Fakultät Mannheim der Universität Heidelberg, Mannheim
- Netherlands (3):
  - Nederlands Kanker Instituut Antoni van Leeuwenhoek, Amsterdam
  - Radboud University Medical Center, Nijmegen
  - Canisius-Wilhelmina Ziekenhuis Nijmegen, Nijmegen
- Inselspital-Universitätsspital Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Harisinghani MG, Barentsz J, Hahn PF, Deserno WM, Tabatabaei S, van de Kaa CH, de la Rosette J, Weissleder R. Noninvasive detection of clinically occult lymph-node metastases in prostate cancer. N Engl J Med. 2003 Jun 19;348(25):2491-9. doi: 10.1056/NEJMoa022749. PMID 12815134
- [Background] Heesakkers RA, Hovels AM, Jager GJ, van den Bosch HC, Witjes JA, Raat HP, Severens JL, Adang EM, van der Kaa CH, Futterer JJ, Barentsz J. MRI with a lymph-node-specific contrast agent as an alternative to CT scan and lymph-node dissection in patients with prostate cancer: a prospective multicohort study. Lancet Oncol. 2008 Sep;9(9):850-6. doi: 10.1016/S1470-2045(08)70203-1. Epub 2008 Aug 15. PMID 18708295
- [Background] Heesakkers RA, Jager GJ, Hovels AM, de Hoop B, van den Bosch HC, Raat F, Witjes JA, Mulders PF, van der Kaa CH, Barentsz JO. Prostate cancer: detection of lymph node metastases outside the routine surgical area with ferumoxtran-10-enhanced MR imaging. Radiology. 2009 May;251(2):408-14. doi: 10.1148/radiol.2512071018. PMID 19401573
- [Background] D'Amico AV, Whittington R, Malkowicz SB, Schultz D, Blank K, Broderick GA, Tomaszewski JE, Renshaw AA, Kaplan I, Beard CJ, Wein A. Biochemical outcome after radical prostatectomy, external beam radiation therapy, or interstitial radiation therapy for clinically localized prostate cancer. JAMA. 1998 Sep 16;280(11):969-74. doi: 10.1001/jama.280.11.969. PMID 9749478